CLINICAL TRIAL: NCT01543568
Title: AflibercepT for Subjects Who Are Incomplete Responders to mUltiple Intravitreal Injections of Ranibizumab, Anti-VegF (The TURF Study)
Brief Title: Study for Recalcitrant Age Related Macular Degeneration
Acronym: TURF
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: David M. Brown, M.D. (Other)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor-Investigator, David M. Brown, M.D., Director of Research, Greater Houston Retina Research
Organization: Greater Houston Retina Research (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TURF-01
Record Dates: First submitted 2012-02-27; First posted 2012-03-05 (Estimated); Results first posted 2017-01-02 (Estimated); Last update posted 2017-01-02 (Estimated); Status verified 2016-11

CONDITIONS: Age Related Macular Degeneration
Keywords: Age related Macular Degeneration; Recalcitrant Age Related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration | interventions — aflibercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 2.0 mg intravitreal Aflibercept (Other): open label, Subjects seen monthly & given mandatory 2.0 mg aflibercept at baseline, months 1, 2 and 4. Pro re nata (PRN) retreatment at months 3 and 5 was performed upon evidence of disease on spectral domain-optical coherence tomography (SD-OCT)
  Interventions: Drug: aflibercept 2.0 mg

INTERVENTIONS:
Drug: aflibercept 2.0 mg — Intravitreal aflibercept injection 2.0 mg
  Other Names: Veg F Trap

SUMMARY:
50 Patients with recalcitrant exudative age-related macular degeneration with a history of retinal or subretinal fluid after multiple intravitreal injections with ranibizumab 0.5mg and subsequently treated with ranibizumab 2.0mg, who are incomplete responders to 2.0mg of ranibizumab.

DETAILED DESCRIPTION:
The rationale for the TURF trial is based on the greater binding affinity of VEGF Trap-eye, which theoretically may prove to be more effective for recalcitrant wet AMD and therefore may demonstrate a positive impact on visual acuity and the foveal anatomy of subjects who have a history of a less than optimal anatomical and visual response to multiple intravitreal injections of 2.0mg (super-dose) ranibizumab. Based on the anatomical data from the VIEW1 and VIEW2 trials, approximately 70% of VEGF-Trap eye patients had no evidence of fluid on OCT compared to approximately 55% of ranibizumab patients. One potential interpretation of this clinical data is that the increased binding affinity and longer half-life of VEGF-Trap eye result in the resolution of more fluid for a longer duration of effect.

Patients to be enrolled in this study have a history of requiring monthly dosing of ranibizumab 2.0mg to achieve maximum resolution of fluid on OCT and increased visual acuity. These patients initially showed minimal fluid resolution visual acuity gains while treated with Lucentis (0.5mg ranibizumab) and were subsequently treated with 2.0mg monthly. It is expected that treating these same patients with 2.0mg EYLEA™ (aflibercept injection for eye) will maintain the fluid resolution on OCT and visual acuity gains previously requiring a super-dose of ranibizumab.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent and comply with study assessments for the full duration of the study
* Age > 50 years
* Choroidal neovascularization secondary to AMD
* History of treatment with 0.5mg ranibizumab followed by 2.0mg ranibizumab for AMD
* Best corrected visual acuity in the study eye between 20/20 to 20/400 using an ETDRS chart

Exclusion Criteria:

* Pregnancy (positive pregnancy test) or lactation
* Premenopausal women not using adequate contraception. The following are considered effective means of contraception: surgical sterilization or use of oral contraceptives, barrier contraception with either a condom or diaphragm in conjunction with spermicidal gel, an IUD, or contraceptive hormone implant or patch.
* Participation in another simultaneous medical investigation or trial
* Prior treatment with anti-VEGF therapy in the study eye within 28 days of baseline
* Prior treatment with PDT within the past 3 months or more than 4 prior PDT treatments.
* Presence of significant subfoveal fibrosis or atrophy.
* Prior treatment with intravitreal aflibercept injection
* Prior treatment with triamcinolone in the study eye within 6 months of BSL.
* Prior treatment with dexamethasone in the study eye within 30 days prior to BSL
* Intraocular surgery (including cataract surgery) in the study eye within 2 months preceding Baseline
* History of vitrectomy surgery, submacular surgery, or other surgical intervention for AMD in the study eye
* Active intraocular inflammation (grade trace or above) in the study eye
* Current vitreous hemorrhage in the study eye
* History of rhegmatogenous retinal detachment or macular hole (Stage 3 or 4) in the study eye
* Active infectious conjunctivitis, keratitis, scleritis, or endophthalmitis in either eye
* Uncontrolled glaucoma in the study eye (defined as IOP ≥ 30 mmHg despite treatment with anti-glaucoma medication)
* History of cerebral vascular accident, myocardial infarction, transient ischemic attacks within 3 months of study enrollment.
* History of allergy to fluorescein, ICG or iodine, not amenable to treatment
* History of retinal pigment epithelial tear or rip

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2012-02; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David M Brown, MD, Principal Investigator — Director Greater Houston Research
Locations (1):
- Retina Consultants of Houston, Houston, Texas, United States

REFERENCES:
- [Background] Aflibercept (eylea) for age-related macular degeneration. Med Lett Drugs Ther. 2012 Feb 6;54(1383):9-10. No abstract available. PMID 22354219
- [Background] Ohr M, Kaiser PK. Intravitreal aflibercept injection for neovascular (wet) age-related macular degeneration. Expert Opin Pharmacother. 2012 Mar;13(4):585-91. doi: 10.1517/14656566.2012.658368. Epub 2012 Feb 3. PMID 22300011
- [Background] Gragoudas ES, Adamis AP, Cunningham ET Jr, Feinsod M, Guyer DR; VEGF Inhibition Study in Ocular Neovascularization Clinical Trial Group. Pegaptanib for neovascular age-related macular degeneration. N Engl J Med. 2004 Dec 30;351(27):2805-16. doi: 10.1056/NEJMoa042760. PMID 15625332
- [Background] CATT Research Group; Martin DF, Maguire MG, Ying GS, Grunwald JE, Fine SL, Jaffe GJ. Ranibizumab and bevacizumab for neovascular age-related macular degeneration. N Engl J Med. 2011 May 19;364(20):1897-908. doi: 10.1056/NEJMoa1102673. Epub 2011 Apr 28. PMID 21526923
- [Background] Rosenfeld PJ, Brown DM, Heier JS, Boyer DS, Kaiser PK, Chung CY, Kim RY; MARINA Study Group. Ranibizumab for neovascular age-related macular degeneration. N Engl J Med. 2006 Oct 5;355(14):1419-31. doi: 10.1056/NEJMoa054481. PMID 17021318
- [Background] Brown DM, Kaiser PK, Michels M, Soubrane G, Heier JS, Kim RY, Sy JP, Schneider S; ANCHOR Study Group. Ranibizumab versus verteporfin for neovascular age-related macular degeneration. N Engl J Med. 2006 Oct 5;355(14):1432-44. doi: 10.1056/NEJMoa062655. PMID 17021319
- [Background] Rosenfeld PJ, Moshfeghi AA, Puliafito CA. Optical coherence tomography findings after an intravitreal injection of bevacizumab (avastin) for neovascular age-related macular degeneration. Ophthalmic Surg Lasers Imaging. 2005 Jul-Aug;36(4):331-5. PMID 16156152
- [Background] Avery RL, Pieramici DJ, Rabena MD, Castellarin AA, Nasir MA, Giust MJ. Intravitreal bevacizumab (Avastin) for neovascular age-related macular degeneration. Ophthalmology. 2006 Mar;113(3):363-372.e5. doi: 10.1016/j.ophtha.2005.11.019. Epub 2006 Feb 3. PMID 16458968
- [Background] Fung AE, Lalwani GA, Rosenfeld PJ, Dubovy SR, Michels S, Feuer WJ, Puliafito CA, Davis JL, Flynn HW Jr, Esquiabro M. An optical coherence tomography-guided, variable dosing regimen with intravitreal ranibizumab (Lucentis) for neovascular age-related macular degeneration. Am J Ophthalmol. 2007 Apr;143(4):566-83. doi: 10.1016/j.ajo.2007.01.028. PMID 17386270
- [Background] Iida T, Yannuzzi LA, Spaide RF, Borodoker N, Carvalho CA, Negrao S. Cystoid macular degeneration in chronic central serous chorioretinopathy. Retina. 2003 Feb;23(1):1-7; quiz 137-8. doi: 10.1097/00006982-200302000-00001. PMID 12652224
- [Background] Imamura Y, Fujiwara T, Spaide RF. Fundus autofluorescence and visual acuity in central serous chorioretinopathy. Ophthalmology. 2011 Apr;118(4):700-5. doi: 10.1016/j.ophtha.2010.08.017. Epub 2010 Nov 5. PMID 21055816
- [Background] Stewart MW, Rosenfeld PJ. Predicted biological activity of intravitreal VEGF Trap. Br J Ophthalmol. 2008 May;92(5):667-8. doi: 10.1136/bjo.2007.134874. Epub 2008 Mar 20. PMID 18356264
- [Background] Kaiser PK. Vascular endothelial growth factor Trap-Eye for diabetic macular oedema. Br J Ophthalmol. 2009 Feb;93(2):135-6. doi: 10.1136/bjo.2008.144071. No abstract available. PMID 19174397
- [Background] Holash J, Davis S, Papadopoulos N, Croll SD, Ho L, Russell M, Boland P, Leidich R, Hylton D, Burova E, Ioffe E, Huang T, Radziejewski C, Bailey K, Fandl JP, Daly T, Wiegand SJ, Yancopoulos GD, Rudge JS. VEGF-Trap: a VEGF blocker with potent antitumor effects. Proc Natl Acad Sci U S A. 2002 Aug 20;99(17):11393-8. doi: 10.1073/pnas.172398299. Epub 2002 Aug 12. PMID 12177445
- [Background] Eyetech Study Group. Preclinical and phase 1A clinical evaluation of an anti-VEGF pegylated aptamer (EYE001) for the treatment of exudative age-related macular degeneration. Retina. 2002 Apr;22(2):143-52. doi: 10.1097/00006982-200204000-00002. PMID 11927845
- [Derived] Wykoff CC, Brown DM, Maldonado ME, Croft DE. Aflibercept treatment for patients with exudative age-related macular degeneration who were incomplete responders to multiple ranibizumab injections (TURF trial). Br J Ophthalmol. 2014 Jul;98(7):951-5. doi: 10.1136/bjophthalmol-2013-304736. Epub 2014 Feb 11. PMID 24518078

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from March 2012 to September 2012. 50 subjects from 1 site of the United States from a medical clinic. Each subject was was over 50 years of age, diagnosed with choroidal neovascularization secondary to AMD, and had a history of treatment with 0.5 mg ranibizumab followed by 2.0 mg ranibizumab for AMD.
Period: Overall Study
Arm/Group | 2.0 mg Intravitreal Aflibercept
Started | 46
Completed | 45
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | 2.0 mg Intravitreal Aflibercept
Number analyzed (Participants) | 46
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 41
Age, Continuous [Mean (Full Range); unit: years] | 77.8 [55 to 95]
Gender [Count of Participants; unit: Participants]
  Female | 24
  Male | 22
Region of Enrollment [Number; unit: participants]
  United States | 46

OUTCOME MEASURES:

1. Primary Outcome: The Number of Patients With no Fluid on OCT
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | 2.0 mg Intravitreal Aflibercept
Number analyzed (Participants) | 46
participants | 10

2. Secondary Outcome: Mean Change in OCT Central Foveal Thickness
Time Frame: 6 Months
Measure: Mean (Full Range); unit: micrometers
Arm/Group | 2.0 mg Intravitreal Aflibercept
Number analyzed (Participants) | 46
micrometers | -27.3 [-381 to 59]

3. Secondary Outcome: Average Time to Resolution of Intraretinal Cysts and Sub Retinal Fluid on OCT
Time Frame: 6 months
Measure: Mean (Full Range); unit: months
Arm/Group | 2.0 mg Intravitreal Aflibercept
Number analyzed (Participants) | 46
months | 4 [0 to 6]

4. Secondary Outcome: The Percentage of Patients Who Lose > 15 Letters Visual Acuity
Time Frame: 6 Months
Measure: Number; unit: Percentage of patients
Arm/Group | 2.0 mg Intravitreal Aflibercept
Number analyzed (Participants) | 46
Percentage of patients | 0

5. Secondary Outcome: Mean Change in Visual Acuity (BCVA)
Description: Change in Early Treatment of Diabetic Retinopathy Study Best Corrected Visual Acuity (ETDRS-BCVA) from baseline to month 6. BCVA is measured using an eye chart and is reported as the number of letters read correctly using the ETDRS Scale (ranging from 0 to 100 letters) in the study eye. The lower the number of letters read correctly on the eye chart, the worse the vision (or visual acuity). An increase in the number of letters read correctly means that vision has improved.
Time Frame: 6 Months
Measure: Mean (Full Range); unit: ETDRS BCVA letters
Arm/Group | 2.0 mg Intravitreal Aflibercept
Number analyzed (Participants) | 46
ETDRS BCVA letters | 0.2 [-10 to 13]

6. Secondary Outcome: Quantitative Change in Area (μ) From Baseline in Choroidal Neovascular Lesion Characteristics/Size as Measured by FA/Fundus Photos
Time Frame: 6 Months
Population: Given lack of visual benefit upon switching to aflibercept (Eylea), such analyses were not performed.
Arm/Group | 2.0 mg Intravitreal Aflibercept
Number analyzed (Participants) | 0

7. Secondary Outcome: Mean Number of 0.2 mg Aflibercept Injections Administered
Time Frame: at 6 months
Measure: Mean (Full Range); unit: injections
Arm/Group | 2.0 mg Intravitreal Aflibercept
Number analyzed (Participants) | 46
injections | 5.6 [4 to 6]

ADVERSE EVENTS:
Arm/Group | 2.0 mg Intravitreal Aflibercept
Serious Adverse Events (participants affected / at risk) | 9/45
Other Adverse Events (participants affected / at risk) | 6/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 2.0 mg Intravitreal Aflibercept (N=45)
Urinary Tract Infection (Infections and infestations) | 2
Death (Cardiac disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 2.0 mg Intravitreal Aflibercept (N=45)
Cataract Progression (Eye disorders) | 3
Geographic atrophy progression (Eye disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes